CLINICAL TRIAL: NCT04970641
Title: Three Good Things (3GT) - Intervention for Transitional Care Patients at the Mayo Clinic Bloomer Critical Access Hospital
Brief Title: Three Good Things (3GT) - Intervention for Transitional Care Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Restrictions to recruitment due to staffing shortages and low patient census
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lori M. Miller, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-003878
Record Dates: First submitted 2021-07-19; First posted 2021-07-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Positive Thinking; Psychology, Positive; Resilience, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3GT journaling group (Experimental): Subjects will participate in the Three Good Things (3GT) Positive Psychology journaling activity daily for six weeks.
  Interventions: Behavioral: Three Good Things (3GT) Positive Psychology journaling activity
- Non-journaling group (No Intervention): Subjects will not participate in the evening journal activity.

INTERVENTIONS:
Behavioral: Three Good Things (3GT) Positive Psychology journaling activity — Evening journaling activity each day to reflect on three good things that the subject has noticed about their day's events.
  Arms: 3GT journaling group

SUMMARY:
Researchers are doing this research study to learn how the Three Good Things (3GT) Positive Psychology journaling activity affects symptoms of stress, depression, resilience, and happiness.

DETAILED DESCRIPTION:
The purpose of this study is to measure, rank and categorize the subject sample of depression, stress, resilience and happiness scores using quantitative surveys. This research aims to learn how a Three Good Things (3GT) journaling activity affects a subject's symptoms of stress, depression, resilience and happiness. The data will allow the project team to gain an in-depth understanding of the impact of the use of resilience strategies from a hospitalized patient's perspective. The project aims to review if there is a correlation between stress, depression, resiliency, and happiness scores to the use of Positive Psychology.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age.
* Current inpatient at the Mayo Clinic Health System Bloomer Hospital, Bloomer, Wisconsin (a Swing Bed Hospital as defined by the Center for Medicare and Medicaid Services (CMS)).
* Able to speak English.
* Able to answer questionnaires.

Exclusion Criteria:

* Individuals < 18 years of age.
* Patient unwilling or unable to provide consent to participate in this research study.
* Patient under guardianship.
* As determined through self-report, patient in active psychosis, active suicidal ideation, active substance abuse meeting criteria for substance use disorders except for nicotine (the exception is patients with a history of substance abuse that have been in remission for at least one full year).
* Patient diagnosed with obsessive-compulsive disorder, active panic disorder with agoraphobia or other phobic disorder, active Post Traumatic Stress Disorder, or active severe personality disorders.
* Patient with previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | Baseline, 6 weeks
  Change in subject perceived stress measured using the self-reported perceived stress scale (PSS). A 10-item questionnaire assessing individuals' appraisal of stress using a scale of 0=never, 4=very often.

SECONDARY OUTCOMES:
Subjective Depression | Baseline, 6 weeks
  Change in subject depression measured using the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R-10).
Subjective Happiness | Baseline, 6 weeks
  Change in subject happiness measured using the self-reported subjective happiness scale (SHS). A 4-item scale of global subjective happiness. Two items ask respondents to characterize themselves using both absolute ratings and ratings relative to peers, whereas the other two items offer brief descriptions of happy and unhappy individuals and ask respondents the extent to which each characterization describes them.
Subjective Resilience | Baseline, 6 weeks
  Change in subject resiliency scores measured by the Connor-Davidson Resilience Scale (CD-RISC 2)

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Miller, MAOM, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System Bloomer Hospital, Bloomer, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers.